CLINICAL TRIAL: NCT06030687
Title: Multiscale RECIPES (Resilient, Equitable, and Circular Innovations With Partnership and Education Synergies) for Sustainable Food Systems (FoodImage 3; FI3) Free-Living
Brief Title: FoodImage 3 Free-Living
Acronym: FI3FL
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Martin, Corby, K., M.D. (Individual)
Responsible Party: Principal Investigator, John Apolzan, Associate Professor-Research, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-045 A
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Waste Management; Food Supply; Climate; Nutrition Sciences

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Free-Living
  Interventions: Other: Ad libitum data collection

INTERVENTIONS:
Other: Ad libitum data collection — Food purchase, prep, eat and toss data

SUMMARY:
Participants will be asked to use the app to capture data on food purchases, food waste that occurs during food preparation, food waste that is present after eating, and food waste from cabinet and refrigerator/freezer clean-outs. During collection of much of the food waste data, participants will record in the app if food waste will be disposed of via composting, disposal, fed to pets, or garbage/landfill. They will also indicate if the food was spoiled, past the expiration date, etc. This will occur for 4-8 days. Participants should perform the prep and eat occasions 4-8 days. The shopping and toss occasions should be completed for at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 18-65 years
* Willing to be recontacted
* Conducts some of the food shopping, food purchasing, and/or food preparation for their household.
* Internet and/or Wi-Fi availability to complete surveys and send images.
* Ownership of an iPhone 9S or later, operable Apple ID, password, and email address that they are willing and able to use to collect data during the study. Subject acknowledges data usage and associated charges are a result of study.
* Willing to complete all study procedures and adhere to study visit timelines -

Exclusion Criteria:

* Refusal or unable to use an iPhone for study related purposes.
* Not willing to adhere to study procedures and study visit timelines.
* PBRC employee
* Any condition or circumstance that in the judgement of the PI could interfere with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Total weight of household food waste | daily during baseline collection
  weight (g)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be requested. The PI will be notified. The proposed research question must be included. All IPD that underlie results in a publication after a DTA with the institution may be requested.